CLINICAL TRIAL: NCT04946474
Title: Clinical Evaluation and Study on the Combination of Disease and Syndrome With General Treatment for Acute Hemorrhagic Stroke
Brief Title: Clinical Evaluation of the Combination of Symptoms and Symptoms With General Treatment for Acute Hemorrhagic Stroke
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2019412
Record Dates: First submitted 2021-06-27; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Acute Hemorrhagic Stroke
MeSH Terms: interventions — xingnaojing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xingnaojing injection + Shuxuetong oral liquid (Experimental): Xingnaojing injection (administered immediately after joining the group, once a day, treatment for 10 days) + Naoxueshu oral liquid treatment (administered on the 4th day of onset, 3 times a day, treatment for 30 days ).
  Interventions: Drug: Xingnaojing injection + Shuxuetong oral liquid
- Placebo group (Placebo Comparator): Xingnaojing injection simulation agent + Naoxueshu oral liquid simulation agent treatment was given.
  Interventions: Drug: Xingnaojing injection + Shuxuetong oral liquid

INTERVENTIONS:
Drug: Xingnaojing injection + Shuxuetong oral liquid — Xingnaojing injection (administered immediately after joining the group, once a day, treatment for 10 days) + Naoxueshu oral liquid treatment (administered on the 4th day of onset, 3 times a day, treatment for 30 days ).

SUMMARY:
Objective To evaluate whether Xingnaojing injection combined with Naoxueshu oral liquid can significantly improve the clinical outcome of patients with intracerebral hemorrhage.

Secondary objectives included to evaluate whether combined application of Xingnaojing injection and Naoxueshu oral liquid can promote hematoma absorption or reduce perihematoma cerebral edema in patients with intracerebral hemorrhage

DETAILED DESCRIPTION:
Objective To evaluate whether Xingnaojing injection combined with Naoxueshu oral liquid can significantly improve the clinical outcome of patients with intracerebral hemorrhage.

Secondary objectives included to evaluate whether combined application of Xingnaojing injection and Naoxueshu oral liquid can promote hematoma absorption or reduce perihematoma cerebral edema in patients with intracerebral hemorrhage Statistical Methods: The main effective outcomes will be based on a generalized linear model and adjusted for associated confounders.

ELIGIBILITY:
Inclusion Criteria:

* ① It meets the diagnostic criteria of primary cerebral hemorrhage.

  * Within 72 hours of onset.

    * National Institutes of Health Stroke Scale (NIHSS) score ≥4 points.

      ④ Glasgow Coma Scale (GCS) score > Eight points.

      ⑤ Age 18-80. Patient or legal representative informed consent, and sign informed consent.

Exclusion Criteria:

* (1) known to Xingnaojing, cerebral hemorrhage or related drug ingredients allergic.

  * The patients with previous stroke history and remaining sequelae affected the outcome assessment, that is, the modified Ranking scale (MRS) score before the onset of stroke was ≥2 points.

    (3) known by amyloid cerebrovascular disease, vascular malformation, aneurysm, blood coagulation dysfunction, anticoagulation and antiplatelet drug treatment, thrombolysis therapy, bleeding after infarction after conversion, haematology, moyamoya disease, primary or metastatic tumor, venous sinus thrombosis, and vascular inflammation caused by clear etiology of patients with cerebral hemorrhage or primary intraventricular hemorrhage.

(Note: "After anticoagulant or antiplatelet therapy" refers to patients with intracerebral hemorrhage following anticoagulant and antiplatelet therapy, and these patients were excluded from this study.) (4) Patients with traumatic cerebral hemorrhage. (5) patients with active gastrointestinal ulcer or other definite tendency of rebleeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
self-care | after 90 days
  90 days of self-care (mRS 0-2 points)

SECONDARY OUTCOMES:
NIHSS | on day 14 of onset
  NIHSS score improvement on day 14 of onset

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Yniversity Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No